CLINICAL TRIAL: NCT06209372
Title: The Efficiency of Preoperative Pericapsular Nerve Group Block Applied With Ultrasound in Patients With Hip Fracture and Its Effect on the Success of Spinal Anesthesia (PENG)
Brief Title: The Efficiency of Preoperative Pericapsular Nerve Group Block Applied With Ultrasound and Success of Spinal Anesthesia
Acronym: PENG
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Eyyup Sabri Ozden, Assistant Professor, Suleyman Demirel University
Other Study IDs: 281570
Record Dates: First submitted 2023-10-05; First posted 2024-01-17 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Efficiency; Spinal Anesthesia; Block
Keywords: Fracture, Hip;; Block, Pericapsular Nerve Group;; Anesthesia, Spinal;; Success;; Ultrasound
MeSH Terms: conditions — Bites and Stings; Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group PENG (P): Group PENG (P) received the PENG block with 20 mL of 0.25% bupivacaine under ultrasound guidance at preoperative care unit (PCU). The linear ultrasound probe for the PENG block was placed parallel to the imaginary line passing between the spina iliaca anterior inferior and the iliopubic eminence (IPE). The 80mm peripheral block needle was advanced with the in-plane technique, and the block was completed by injecting 20 mL of 0.25% bupivacaine.
  Interventions: Procedure: Group PENG
- Group Control (C): Group Control (C), patients who did not prefer the block were given 10 mg of IV bolus tramadol, followed by 10 mg/hr infusion at preoperative care unit (PCU).
  Interventions: Drug: Group C

INTERVENTIONS:
Procedure: Group PENG — Pericapsular Nerve Group Block (PENG)
  Groups: Group PENG (P)
Drug: Group C — Tramadol infusion
  Groups: Group Control (C)

SUMMARY:
We aimed to investigate the effectiveness of the pericapsular nerve group (PENG) block applied with preoperative ultrasonography (USG) in patients who were operated on under spinal anesthesia due to hip fracture and whether it influences spinal anesthesia success. The files of 100 patients were reviewed observationally, and 60 patients were included in the study. The patients were divided into two groups: Group P (n = 30) comprising patients who underwent PENG block under USG guidance before the start of surgery and the control group (Group C; n = 30) of patients in whom tramadol infusion was started. From the files of the patients, the transition from the bed to the operating table, lateral decubitus position, skin incision, postoperative exit, postoperative 2nd, 4th, 12th, and 24th hour numeric rating scale (NRS) values, spinal anesthesia duration and number of attempts, and perioperative total tramadol consumption were recorded. During the transfer from the patient bed to the operating table and during the lateral decubitus position, postoperative exit and postoperative 2nd, 4th, 8th, 12th, and 24th hour NRS values were found to be significantly lower in Group P. In addition, lower spinal anesthesia time, lower number of spinal anesthesia attempts, and lower perioperative total tramadol consumption were detected in Group P. We found that PENG block applied preoperatively to patients with spinal anesthesia decreased the perioperative pain score, increased the success of spinal anesthesia by facilitating positioning for spinal anesthesia, and decreased the need for postoperative opioids.

DETAILED DESCRIPTION:
This study was conducted after obtaining approval from the Clinical Research Ethics Committee of Süleyman Demirel University (SDU) Faculty of Medicine (Decision no. 281570, dated 10.06.2022). Between December 2021 and June 2022, hip fracture surgery was performed on 100 patients 18 yr and older who were in the American Society of Anesthesiologists' (ASA) I-II-III risk group, using spinal anesthesia at the SDU Faculty of Medicine Hospital Operating Room. The patients' files were reviewed, including those who received the PENG block ın the PCU and those who did not.

Patients with a history of chronic pain, previous hip joint surgery, those who had an unsuccessful PENG block application, and those with missing data in their medical records were excluded from the study (Figure 1). After excluding patients who did not meet the study criteria, 60 patients, including 30 who received the PENG block and 30 who did not, were included in the study.

When the patients were brought to the PCU, they were informed about the procedure, and written consent was obtained after explanation. Standard ASA monitoring was performed after obtaining consent. Patients with full cooperation were informed about the numeric rating scale (NRS), and their pain scores were recorded on the pain follow-up form. If there were no contraindications, 1 g of paracetamol was administered to all patients. After the pain score was assessed in the PCU, a preemptive PENG block was applied, or 10 mg of tramadol IV push was administered, followed by 10 mg/hr infusion, depending on the patient's clinical condition. Group PENG (P) received the PENG block with 20 mL of 0.25% bupivacaine under ultrasound guidance at PCU. The linear USG probe for the PENG block was placed parallel to the imaginary line passing between the spina iliaca anterior inferior and the iliopubic eminence (IPE). The 80mm peripheral block needle was advanced with the in-plane technique, and the block was completed by injecting 20 mL of 0.25% bupivacaine. In Group Control (C), patients who did not prefer the block were given 10 mg of IV bolus tramadol, followed by 10 mg/hr infusion at PCU.

The NRS scores of all patients were recorded, and if the NRS score was >3, 10 mg of IV bolus tramadol was administered with a waiting time of 30 min before starting the surgical intervention. After 30 min of analgesic treatment, the patient was transported to the operating table.

If regional anesthesia was planned for patients, except for specific situations, unilateral hypobaric spinal anesthesia was applied in the standard lateral decubitus position. All patients were administered 1.5 mL of 0.5% bupivacaine (7.5 mg) + 1.5mL of distilled water + 0.25 mL of fentanyl (12.5 mcg) prepared with a 25 G - 90 mm cutting-edge disposable spinal needle. The number of attempts, the success of the dural puncture, and the time of skin incision were recorded on the anesthesia follow-up form. In addition, the level of spinal anesthesia was determined by the pinprick test at the 5th min.

The patients' demographic data, the surgical procedure and duration, the patient's postoperative discharge site, heart rate, mean arterial pressure (MAP), and peripheral saturation (SpO2) values measured during pre-analgesic application 30 min after, before spinal anesthesia, during skin incision, during the first hour of surgery, and postoperative discharge were recorded and evaluated from hospital information system data, anesthesia follow-up forms, surgical notes, perioperative pain monitoring forms, and discharge reports. Similarly, the spinal anesthesia duration (the time between the start of spinal anesthesia to skin incision), the number of spinal anesthesia attempts, the patient's position during the transfer from the bed to the operating table, the lateral decubitus position, skin incision, and NRS values at postoperative exit, and at the 2nd, 4th, 12th, and 24th hr postoperatively were recorded and evaluated. In the same manner, the total amount of tramadol administered during and after surgery, and postoperative complications (postoperative nausea and vomiting, hypotension, quadriceps muscle weakness, infection, hematoma, local anesthetic toxicity) were recorded and evaluated.

Statistical Analysis This article describes a statistical analysis performed on data using the Statistical Package for Social Science (SPSS) version 24. Qualitative data was presented as numbers and percentages, while quantitative data was presented as means and standard deviations (SD). The Kolmogorov-Smirnov and Shapiro-Wilk tests were used to check for normal distribution of continuous variables. The student's t-test was used to compare two independent groups of normally distributed variables, the Mann Whitney U test was used to compare two independent groups of variables that did not have a normal distribution, and the chi-square test was used to compare categorical data.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* American Society of Anesthesiologists' (ASA) I-II-III

Exclusion Criteria:

* Patients with a history of chronic pain,
* Previous hip joint surgery,
* Unsuccessful PENG block or spinal anesthesia application,
* Missing data in their records
* History of bleeding diathesis
* Increased intracranial pressure
* Severe mitral and/or aortic stenosis
* Allergic to the medications used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hip fracture surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in pain score after applying Pericapsular Nerve Group Block (PENG) | 30 minutes after applying PENG block
  In line with the literature, we determined that the NRS value significantly decreased during positioning for spinal anesthesia in the group where the PENG block was applied.
Pericapsular Nerve Group Block (PENG) block facilitates the success of spinal anesthesia | 30 minutes after applying PENG block
  Effective pain control facilitates the success of spinal anesthesia by making positioning and application easier is supported by our study.

CONTACTS AND LOCATIONS:
Overall Officials: Eyyup Ozden, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Hospital, Isparta, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Acharya U, Lamsal R. Pericapsular Nerve Group Block: An Excellent Option for Analgesia for Positional Pain in Hip Fractures. Case Rep Anesthesiol. 2020 Mar 12;2020:1830136. doi: 10.1155/2020/1830136. eCollection 2020. PMID 32231802
- [Result] Afolayan JM, Areo PO, Adegun PT, Ogundipe KO, Filani AB. Comparison of ease of induction of spinal anaesthesia in sitting with legs parallel on the table versus traditional sitting position. Pan Afr Med J. 2017 Nov 13;28:223. doi: 10.11604/pamj.2017.28.223.6992. eCollection 2017. PMID 29629009